CLINICAL TRIAL: NCT05753748
Title: A Multicenter Randomized Controlled Trial of Surveillance vs. Endoscopic Therapy for Barrett's Esophagus With Low-grade Dysplasia (The SURVENT Trial)
Brief Title: Surveillance vs. Endoscopic Therapy for Barrett's Esophagus With Low-grade Dysplasia
Acronym: SURVENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Baylor University (Other); University of North Carolina (Other); Medical University of South Carolina (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-4972.cc; NCI-2023-00787 (Other: CTRP); 1U34DK124174-01 (NIH)
Record Dates: First submitted 2023-01-23; First posted 2023-03-03 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Barretts Esophagus With Dysplasia; Barrett Esophagus; Esophageal Adenocarcinoma
Keywords: Barrett Esophagus; Esophageal Adenocarcinoma; Dysplasia
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endoscopic Surveillance (No Intervention): Subjects in the randomized control trial and observational cohort study, undergoing surveillance endoscopy will undergo surveillance biopsies in a 4-quadrant fashion every 1 cm throughout the extent of the Barrett's esophagus using the Seattle biopsy protocol, along with targeted biopsies from any visible lesions. For incident low grade dysplasia (newly diagnosed low grade dysplasia - within 12 months of enrollment), surveillance endoscopies will be performed every 6 months for the first year and then annually until the end of the study period. For prevalent low grade dysplasia (diagnosed >1 year prior to enrollment), surveillance endoscopies will be performed annually until the end of the study period. The number of evaluations will depend on a subject's enrollment time.
- Endoscopic Eradication Therapy (Experimental): Subjects undergoing endoscopic eradication therapy will undergo radiofrequency ablation every 2-3 months until complete eradication of intestinal metaplasia (CE-IM) is achieved or 5 treatments have been delivered, whichever is first. After achieving CE-IM, surveillance endoscopy will performed every 6 months for the first year and annually thereafter until the end of the study period. Surveillance biopsies will be obtained using a standardized protocol.
  Interventions: Procedure: Endoscopic Eradication Therapy

INTERVENTIONS:
Procedure: Endoscopic Eradication Therapy — Endoscopic eradication therapy is a procedure performed to destroy the precancerous cells at the bottom of your esophagus, so that healthy cells can grow in their place. It involves procedures to either remove precancerous tissue or burn it. These procedures are performed through the endoscope.
  Arms: Endoscopic Eradication Therapy

SUMMARY:
The purpose of this study is to learn the best approach to treating patients with known or suspected Barrett's esophagus by comparing endoscopic surveillance to endoscopic eradication therapy.

To diagnose and manage Barrett's esophagus and low-grade dysplasia, doctors commonly use procedures called endoscopic surveillance and endoscopic eradication therapy. Endoscopic surveillance is a type of procedure where a physician will run a tube with a light and a camera on the end of it down the patients throat and remove a small piece of tissue. The piece of tissue, called a biopsy, is about the size of the tip of a ball-point pen and is checked for abnormal cells and cancer cells.

Endoscopic eradication therapy is a kind of surgery which is performed to destroy the precancerous cells at the bottom of the esophagus, so that healthy cells can grow in their place. It involves procedures to either remove precancerous tissue or burn it. These procedures can have side effects, so it is not certain whether risking those side effects is worth the benefit people get from the treatments.

While both of these procedures are widely accepted approaches to managing the condition, there is not enough research to show if one is better than the other.

Barrett's esophagus and low-grade dysplasia does not always worsen to high-grade dysplasia and/or cancer. In fact, it usually does not. So, if a patient's dysplasia is not worsening, doctors would rather not put patients at risk unnecessarily. On the other hand, endoscopic eradication therapy could possibly prevent the worsening of low-grade dysplasia into high-grade dysplasia or cancer (esophageal adenocarcinoma) in some patients. Researchers believe that the results of this study will help doctors choose the safest and most effective procedure for their patients with Barrett's esophagus and low-grade dysplasia.

This is a multicenter study involving several academic, community and private hospitals around the United States. Up to 530 participants will be randomized. This study will also include a prospective observational cohort study of up to 150 Barrett's esophagus and low grade dysplasia patients who decline randomization in the randomized control trial but undergo endoscopic surveillance (Cohort 1) or endoscopic eradication therapy (Cohort 2), and are willing to provide longitudinal observational data.

DETAILED DESCRIPTION:
Methodology:

Patients with Barrett's esophagus and low grade dysplasia will be recruited in the multicenter trial. Patients will be randomized into endoscopic eradication therapy or endoscopic surveillance.

Subjects in the randomized control trial and observational cohort study, undergoing surveillance endoscopy will undergo surveillance biopsies in a 4-quadrant fashion every 1 cm throughout the extent of the Barrett's Esophagus using the Seattle biopsy protocol, along with targeted biopsies from any visible lesions. For incident low grade dysplasia (newly diagnosed low grade dysplasia - within 12 months of enrollment), surveillance endoscopies will be performed every 6 months for the first year and then annually until the end of the study period. For prevalent low grade dysplasia (diagnosed >1 year prior to enrollment), surveillance endoscopies will be performed annually until the end of the study period. The number of evaluations will depend on a subject's enrollment time with a maximum follow up period of 4years.

Subjects undergoing endoscopic eradication therapy will undergo radiofrequency ablation every 2-3 months until complete eradication of intestinal metaplasia (CE-IM) is achieved or 5 treatments have been delivered, whichever is first. After achieving CE-IM, surveillance endoscopy will performed every 6 months for the first year and annually thereafter until the end of the study period. Surveillance biopsies will be obtained using a standardized protocol.

Subjects will be contacted 48-72 hours and 30 days post procedure. All subjects will also receive follow-up phone calls on a semi-annual basis by a blinded central study coordinator.

Study Centers:

To maximize the generalizability of results, this randomized controlled trial will be conducted across different practice settings that include tertiary care centers, closed healthcare networks and large community practices at approximately 21 sites.

Anticipated Number of Participants:

680

* Randomized Control Trial: 530 subjects (265 per study arm)
* Observational: 150 subjects (Cohort 1, n=100 and Cohort 2 n=50)

Statistical Methodology:

Sample size and power calculations were performed for the primary endpoint using a time-to-event analysis. Estimates from available published data were used to approximate the expected progression rates in each arm of the trial. Based on previous clinical trials using similar methodology to confirm diagnosis of low grade dysplasia by expert pathology review, the team estimates 15% of patients with low grade dysplasia would progress to the composite primary endpoint in the surveillance arm compared to 6% in the endoscopic eradication therapy arm. T plan to accrue subjects for 3.5 years and follow them over time and record their time until progression to the primary endpoint or their censoring time if they do not progress. Follow-up observation will continue for approximately 1 year after the last subject is enrolled. Using this term of follow-up and assuming an exponential survival curve in each group and one interim analysis for efficacy and futility, 213 subjects are needed for analysis in each group to achieve 80% power using a two-sided 0.05 alpha level. Thus, accounting for a 10% non-adherence rate (attrition, subject cross-over) the team plans to enroll and randomize a total of 530 subjects (265 per study arm) who meet the eligibility criteria. A conservative rate of progression has been utilized for this sample size calculation given the significant heterogeneity in progression rates in the published literature. Recognizing that sample size estimation is based on assumptions and if the assumed event rate is lower than expected, there may be a decrease in power. To reduce the likelihood of an underpowered study due to incorrect assumptions, it is proposed to conduct a blinded sample size re-estimation once approximately 40% of the required events are reached.

All randomized subjects who are not identified at the index endoscopy with high grade dysplasia or post-endoscopy esophageal adenocarcinoma are defined as the intention to treat (ITT) population. The time to progression will be calculated from the time of randomization until the endoscopy date on which high grade dysplasia/mucosal post-endoscopy esophageal adenocarcinoma/invasive post-endoscopy esophageal adenocarcinoma is detected. If progression never occurs then the total time the subject is followed will be used as a censoring time. Time until censoring or progression to the primary endpoint of surveillance versus endoscopic eradication therapy will be compared by a log-rank test if the proportional hazards assumption is not violated. The continuous measures of Barrett's esophagus length will be included in the primary model as an independent variable. For all pre-specified analyses, a final two-sided p<0.05 will indicate statistical significance. This study is powered to test the primary hypothesis. However, it also offers the opportunity to conduct several analyses addressing other important patient outcomes. Analyses will be conducted to identify risk factors of progression, as well as factors associated with subsequent absence of low grade dysplasia during follow-up using logistic regression analyses. Potential confounding baseline variables, such as demographics, presence of visible lesions, confirmed low grade dysplasia, multifocal low grade dysplasia, and center differences, will be examined.

ELIGIBILITY:
Inclusion Criteria: Any patient with Barrett's esophagus and low grade dysplasia who provides informed consent AND:

Meets all the following criteria will be eligible for enrollment:

1. Male or female, age ≥18 years,
2. Subject has endoscopic evidence of Barrett's esophagus characterized by the presence of salmon-colored mucosa in the tubular esophagus of at least 1 cm in length as well as endoscopic biopsies from the involved areas demonstrating columnar metaplasia with goblet cells. This inclusion criterion will exclude patients with intestinal metaplasia with dysplasia of the gastric cardia,
3. Biopsies within the previous 12 months demonstrating Barrett's esophagus and low grade dysplasia,
4. Confirmation of low grade dysplasia by expert central pathology panel from biopsies obtained within the previous 12 months (including those obtained from the referring physician),
5. Demonstrated ability to tolerate proton pump inhibitor (PPI) therapy based on patient self-report, and, Ability to discontinue antiplatelet and anticoagulant therapy based on standard guideline recommendations prior to and after endoscopic procedures.

Exclusion Criteria:

1. Pregnancy;
2. Prior endoscopic eradication therapy for Barrett's esophagus;
3. History of high grade dysplasia or post-endoscopy esophageal adenocarcinoma;
4. History of esophageal resection/esophagectomy
5. Active erosive esophagitis (Los Angeles Grade B or higher) - patients are eligible upon resolution of erosive esophagitis;
6. Esophageal strictures precluding passage of the endoscope or treatment catheters - patients are eligible upon resolution of esophageal stricture due to endoscopic dilation or resolution with medical therapy;
7. Esophageal varices or known portal hypertension; and
8. Life expectancy of <2 years as judged by the site investigator. * Presence of a visible lesion (nodularity) at the index endoscopy is not an exclusion criterion. Subjects with visible lesions will undergo endoscopic mucosal resection (EMR) to determine pathology; those with high grade dysplasia or post-endoscopy esophageal adenocarcinoma pathology will exit the study after a 30-day safety follow up.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Neoplastic Progression | Baseline, through study completion
  The occurrence of high grade dysplasia/mucosal post-endoscopy esophageal adenocarcinoma/invasive post-endoscopy esophageal adenocarcinoma at any time during the study period following enrollment.

SECONDARY OUTCOMES:
Work Productivity and Activity | Baseline, through study completion
  The Work Productivity and Activity Index (WPAI) is a 6-item questionnaire that has been adapted to address the impact of reflux symptoms on work and activity burden.
  Patient-centered outcomes (PCOs) have been defined and prioritized by key stakeholders (patients, caregivers, clinicians) and will be compared in Barrett's esophagus patients with low grade dysplasia treated with endoscopic eradication therapy to those undergoing surveillance.
Biomarker Utility | Baseline, through study completion
  Three biomarkers of interest (p53, TissueCypher and WATS3D) will be collected to examine the relationship between biomarker results and the primary efficacy outcome.
Esophageal Adenocarcinoma (EAC) progression rate | Baseline, through study completion
  The proportion of subjects that progress to a diagnosis of invasive post-endoscopy esophageal adenocarcinoma alone during follow up
Patient-Reported Depression, Anxiety, and Gastrointestinal Symptoms | Baseline, through study completion
  NIH PROMIS measures (fixed, short-forms) will be used to measure the following constructs: Depression (4 items), Anxiety (8 items), Gastrointestinal Symptoms (13 items dedicated to GERD) and Global Health (10 items).
  Patient-centered outcomes (PCOs) have been defined and prioritized by key stakeholders (patients, caregivers, clinicians) and will be compared in Barrett's esophagus patients with low grade dysplasia treated with endoscopic eradication therapy to those undergoing surveillance.
Patient-Reported Gastroesophageal Reflux | Baseline, through study completion
  The Gastroesophageal Reflux Questionnaire (GERD-Q; 6 items) will assess severity of reflux symptoms including chest pain, burning, and regurgitation.
  Patient-centered outcomes (PCOs) have been defined and prioritized by key stakeholders (patients, caregivers, clinicians) and will be compared in Barrett's esophagus patients with low grade dysplasia treated with endoscopic eradication therapy to those undergoing surveillance.

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Wani, MD, Principal Investigator — University of Colorado, Denver; Nicholas J Shaheen, MD, MPH, Principal Investigator — University of North Carolina; Valerie Durkalski, MPH, PhD, Principal Investigator — Medical University of South Carolina; Rhonda Souza, MD, Principal Investigator — Baylor University
Locations (23):
- United States (23):
  - University of California, Los Angeles, Los Angeles, California
  - Kaiser Permanente Oakland Medical Center, Oakland, California
  - Kaiser Permanente, San Jose, California
  - University of Colorado, Aurora, Colorado
  - Florida Digestive Health Specialists, Sarasota, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana
  - Johns Hopkins Universtiy, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Long Island Jewish Medical Center, Manhasset, New York
  - Columbia Universtiy, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina
  - University Hospitals Cleveland Medical Center Case Western University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylania, Perelman School of Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas